CLINICAL TRIAL: NCT03090971
Title: Clinical Assessment of the Use of Topical Liquid Diclofenac Following Laser Microporation of Cutaneous Neurofibromas in Patients With Neurofibromatosis Type 1
Brief Title: Use of Topical Liquid Diclofenac Following Laser Microporation of Cutaneous Neurofibromas in Patients With NF1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundação Educacional Serra dos Órgãos (Other)
Responsible Party: Principal Investigator, Mauro Geller, Professor & Chairman of Immunology and Microbiology, Fundação Educacional Serra dos Órgãos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NX101-02-2016
Record Dates: First submitted 2017-03-08; First posted 2017-03-27 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Neurofibromatosis 1; Cutaneous Neurofibroma
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Diclofenac; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cutaneous neurofibromas (Experimental): Each subject will have two treatment neurofibromas and two control neurofibromas. Following microporation, the two treatment neurofibromas will be treated with topical diclofenac while the two control neurofibromas will be treated with topical saline.
  Interventions: Drug: Diclofenac Sodium; Drug: Saline Solution

INTERVENTIONS:
Drug: Diclofenac Sodium — Following microporation, treatment neurofibromas will receive treatment with topical diclofenac
Drug: Saline Solution — Following microporation, control neurofibromas will receive treatment with topical saline

SUMMARY:
This is an open, controlled, prospective, proof-of-concept study, in 7 patients presenting NF1 and cutaneous neurofibromas. This study will include three treatment visits to the study center and three follow-up visits. Treatment will consist of two stages: neurofibroma microporation using the laser device, followed by topical application of one drop of diclofenac 25mg/ml on the surface of the neurofibroma; followed by re-application of one drop of diclofenac, twice daily, for three days. The applications subsequent to the first application will be performed by the patients. Subjects will return to the study center at three day intervals (Assessments 2 & 3) for new microporation and topical diclofenac application, followed by at-home topical diclofenac application for three more days. Assessment 4 will take place 3 days after Assessment 3. Assessment 5 will take place 7 days after the end of the treatment period and Assessment 6 at 30 days after the last application of study drug. The primary efficacy variable in this study is the inflammatory process with the presence of tissue necrosis. The primary safety variable is the occurrence of adverse events considered to be associated with the study drug, occurring during the treatment period.

DETAILED DESCRIPTION:
Neurofibromatosis type 1 (NF1) is an autosomal dominant neurocutaneous syndrome with highly variable clinical manifestations and that has a worldwide incidence of approximately 1/2500. The most common lesion is the cutaneous neurofibroma, appearing on the skin of 90% of adults with NF1. The number of cutaneous neurofibromas in an affected individual can vary from a few to several thousand. These lesions may be surgically removed, but typically recur, and surgical removal often leads to scarring. Intralesional administration of diclofenac was previously reported with favorable results, and significant inflammatory processes were observed within the treated neurofibromas, with tissue necrosis and detachment of some treated neurofibromas, effects that were not observed among the control neurofibromas. The primary objective of this study is to evaluate the use of topical diclofenac in the treatment of cutaneous neurofibromas in patients with NF1. The secondary objective of this study is to assess the safety of the use of topical diclofenac in the treatment of cutaneous neurofibromas in patients with NF1. This is an open, controlled, prospective, proof-of-concept study, in 7 patients presenting NF1 and cutaneous neurofibromas. This study will include three treatment visits to the study center and three follow-up visits. Treatment will consist of two stages: neurofibroma microporation using the laser device, followed by topical application of one drop of diclofenac 25mg/ml on the surface of the neurofibroma; followed by re-application of one drop of diclofenac, twice daily, for three days. The applications subsequent to the first application will be performed by the patients. Subjects will return to the study center at three day intervals (Assessments 2 & 3) for new microporation and topical diclofenac application, followed by at-home topical diclofenac application for three more days. Assessment 4 will take place 3 days after Assessment 3. Assessment 5 will take place 7 days after the end of the treatment period and Assessment 6 30 days after the last application of study drug. The primary efficacy variable in this study is the inflammatory process with the presence of tissue necrosis. The primary safety variable is the occurrence of adverse events considered to be associated with the study drug, occurring during the treatment period. Prior to any study-related procedure, written informed consent will be obtained from the participant. The Clinical Research From will be filled, stored, coded, and the data will be analyzed using GraphPad Prism, v. 5.0. Frequency tables will be generated and central tendencies calculated (mean, median, mode).

ELIGIBILITY:
Inclusion Criteria:

* Adults of both genders, between the ages of 18 and 65;
* NF1, diagnosed clinically by a neurologist, dermatologist, or other specialist knowledgeable about the disease, and defined as:

A known mutation in the gene coding for neurofibromin

or, the presence of 2 of the following 7 clinical manifestations of NF1:

* ≥ 6 café-au-lait macules on the body with diameters greater than 15mm in the greatest diameter;
* two or more neurofibromas of any type or one plexiform neurofibroma
* inguinal or axillary freckling
* two or more Lisch nodules (iris hamartomas)
* optic glioma
* a distinct osseous lesion, such as sphenoid wing dysplasia, pseudoarthrosis of the tibia, macrocephaly, or scoliosis
* a first-degree relative with NF1
* Presence of 4 or more cutaneous neurofibromas measuring 0.5-1.2cm in greatest diameter, present on thorax/abdomen or upper or lower limbs;
* If a woman of childbearing potential, is willing to use a medically acceptable form of contraception (in the judgment of the investigator) for the duration of the study;
* Is able to understand the informed consent form describing the risks of this study, and voluntarily signs the informed consent document;
* Is able to understand and comply with the requirements of the protocol.

Exclusion Criteria:

* Surgical, medical, or investigative treatment for any of the 6 target cutaneous neurofibromas to be evaluated in the study within three months prior to the baseline visit;
* Active infection (bacterial, viral, or fungal) requiring systemic antibiotics within two weeks of the baseline visit;
* Pregnancy or breastfeeding;
* Immunocompromised because of a medical condition;
* Known hypersensitivity to diclofenac or any other NSAID;
* Known hypersensitivity to aspirin;
* has a known hypersensitivity to mannitol, sodium metabisulphite, benzyl alcohol, or propylene glycol;
* Known hypersensitivity to lidocaine;
* Currently receiving or has received with 2 weeks of screening an NSAID (including diclofenac), a COX-2 inhibitor, cyclosporine, methotrexate, an oral anti-diabetic, lithium, digoxin, diuretics, anticoagulants (such as warfarin), or a quinolone antibiotic; except for intralesional diclofenac, these medications will not be allowed during the study; low-dose aspirin used for cardioprotective effects will be allowed;
* Any history of hepatic (including hepatic porphyria) or renal disease resulting in ongoing compromised hepatic or renal function;
* History of a bleeding/coagulation disorder;
* History of gastrointestinal (gastric or intestinal) ulcer disease, Crohn's disease, or ulcerative colitis;
* Laboratory examination at screening that reveals in the opinion of the investigator significant, unstable, and/or untreated renal, hepatic, or metabolic disease/dysfunction;
* White blood cell count at screening that is less than 3000, or a platelet count at screening that is less than 150,000;
* Laboratory evaluation at screening that shows the hemoglobin lower than the lower limit of normal for the laboratory utilized;
* Under treatment for a medical condition that, in the opinion of the investigator, may interfere with the safety of the experimental treatment or with the evaluation of efficacy, including but not limited to cardiovascular and/or respiratory disease;
* Subject is not, in the opinion of the investigator, capable of giving informed consent to participate in the study;
* Subject has received an investigational therapy or procedure for any reason within 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy - presence of inflammatory process in the treated neurofibromas | Throughout the 7-day treatment period and subsequent 30-day follow-up period
  Inflammatory process (redness, exculceration)

SECONDARY OUTCOMES:
Efficacy - presence of tissue necrosis in treated neurofibromas | Throughout the 7-day treatment period and subsequent 30-day follow-up period
  Presence of tissue necrosis in treated neurofibromas
Efficacy - neurofibroma size | Throughout the 7-day treatment period and subsequent 30-day follow-up period
  Reduction in neurofibroma size
Efficacy - neurofibroma detatchment | Throughout the 7-day treatment period and subsequent 30-day follow-up period
  Detachment of the treated neurofibroma
Safety - Adverse events | Throughout the 7-day treatment period and subsequent 30-day follow-up period
  Occurrence of adverse events considered to be associated with the study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Fundação Educacional Serra dos Órgãos - UNIFESO, Teresópolis, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveira LB, Geller M, Cunha KS, Santos A, Bernacchi A, Rubenstein AE, Takirambudde S, Mezitis S, de Almeida Ito Brum C, Darrigo LG Jr, Ribeiro MG. Clinical assessment of the use of topical liquid diclofenac following laser microporation of cutaneous neurofibromas in individuals with neurofibromatosis type 1. Heliyon. 2021 Mar 17;7(3):e06518. doi: 10.1016/j.heliyon.2021.e06518. eCollection 2021 Mar. PMID 33817379